CLINICAL TRIAL: NCT07176026
Title: Follow-Up of Ureteral Stones ≤4 mm: Evaluate the Proportion of Spontaneous Passage and Assess if Symptoms and Stone Characteristics Can Predict Stone Passage
Brief Title: Follow-Up of Ureteral Stones ≤4 mm
Status: Enrolling by invitation | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-04897-01
Record Dates: First submitted 2025-06-03; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Biospecimen Retention: Samples Without DNA — S-creatinine, blood test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Follow-up with S-creatine, questionnaire and CT

SUMMARY:
The goal of this clinical trial is to evaluate the proportion of ureteral stones ≤4 mm that pass spontaneously within 4 and 8 weeks and assess if pain, blood test (S-creatinine), stone size, stone location and hydronephrosis can predict stone passage. The participants will be asked to fill in a questionare regarding symptoms, give a blood test and undergo a follow-up computed tomography.

DETAILED DESCRIPTION:
All patients with a diagnosis of ureteral stone ≤4 mm at the Emergency Department in Helsingborg will be asked to participate. If they give consent data regarding age, gender, stone size, stone location, hydronephrosis, S-creatinine, treatments and results from the follow up CT is extraced from the medical records.

ELIGIBILITY:
Inclusion Criteria:

* all patients with acute renal colic where a CT within 24 hours shows an ureteral stone ≤ 4mm and there is no need for acute intervention.

Exclusion Criteria:

* Those who decline to participate, those who are put under guardianship or is less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with acute renal colic where a CT within 24 hours shows a ureteral stone ≤ 4mm.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of ureteral stones ≤ 4mm that pass spontaneously | From enrolement to passage of the stone or maximum 8 weeks.
Number of participants with residual pain | From enrolement to passage of the stone or maximum 8 weeks.
  Residual pain is measured with VAS (visual analogue scale), values 0-10. VAS 0 = no pain and VAS 10 = worst possible pain.

SECONDARY OUTCOMES:
QoL form including sick leave and return to full ADL | From enrolement to passage of the stone or maximum 8 weeks.
  Questionnaire specifically designed for this study, including questions about pain (regarding pain: how often, how severe/ VAS, need for pain medication) and the ability/ inability to work as usual. VAS: visual analougus scale 0-10, 0 = no pain and 10 = worst possible pain.
Proportion of ureteral stone that have passed according to anatomical localisation, S-creatinine and presence of hydronephrosis. | From enrolement to passage of the stone or maximum 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Wagenius, PhD, Principal Investigator — University of Lund
Locations (2):
- Sweden (2):
  - Department of Urology, Helsingborg
  - Department of Urology, KI Huddinge, Stockholm

IPD SHARING:
Plan to Share IPD: No